CLINICAL TRIAL: NCT04852055
Title: Effect of an Advance Care Planning Intervention on Documentation of Advance Directives and Goals of Care in Assisted Living Centers
Brief Title: Effect of an Advance Care Planning Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Vincent Mor, Florence Pirce Grant University Professor, Professor of Health, Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2008002779; 3U54AG063546-02S1 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2023-09-11 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-09

CONDITIONS: Dementia
Keywords: assisted living facilities; dementia; advance care planning
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Patients and proxies in assisted living centers randomized to the usual care arm have advance care planning discussions with a clinician at admission, annually, and sometimes with a hospitalization or other change in condition. There is no standardized decision- or conversation-support tools used to have these discussions.
- Information (Experimental): Patients and proxies in assisted living centers randomized to the information arm will receive a letter from their clinician with a link to an educational video describing the goals of care and how specific treatment decisions align with these goals. Patients and proxies will also continue to receive usual care advance care planning conversations.
  Interventions: Behavioral: Advance Care Planning Video

INTERVENTIONS:
Behavioral: Advance Care Planning Video — Clinical assistants determine who is the correct person to receive the informational materials. If the patient is the correct recipient, clinicians will send the informational materials to the patient at the assisted living center. If the proxy is the correct recipient, the clinical assistant will determine whether or not the proxy is using the existing online portal. If the proxy is using the portal, the informational materials will be sent electronically. If the proxy does not access the portal, the informational materials will be sent to their residences.
  Arms: Information

SUMMARY:
The intervention being studied is an advance care planning intervention. The trial has two arms: usual care and information arm.

DETAILED DESCRIPTION:
Eligible patients whose assisted living centers are randomized to the information arm will receive a letter from their clinician with links to informational video. Eligible patients whose assisted living centers are randomized to the usual care arm have advance care planning discussions with a clinician at admission, annually, and sometimes with a hospitalization or other change in condition.

ELIGIBILITY:
Inclusion Criteria:

* Partnering assisted living center with at least 20 patients with a dementia diagnosis (based on International Classification of Diseases, version 10 codes)
* Patients not on hospice
* Patients who do not have comfort care or do-not-hospitalize orders at baseline

Exclusion Criteria:

* Partnering assisted living center with less than 20 patients with a dementia diagnosis (based on International Classification of Diseases, version 10 codes)
* Patients on hospice
* Patients with comfort care or do-not-hospitalize orders at baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2364 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mor, PhD, Principal Investigator — Brown University, School of Public Health
Locations (1):
- Bluestone Physician Services, Stillwater, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Assisted Living Centers
Period: Overall Study
Arm/Group | Usual Care | Information
Started | 1166; 80 Assisted Living Centers | 1198; 80 Assisted Living Centers
Completed | 997; 79 Assisted Living Centers | 1011; 80 Assisted Living Centers
Not Completed | 169; 1 Assisted Living Centers | 187; 0 Assisted Living Centers

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Information | Total
Number analyzed (Participants) | 997 | 1011 | 2008
Age, Continuous [Mean (Standard Deviation); unit: years] | 83.0 (7.5) | 83.1 (7.6) | 83.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 695 | 707 | 1402
  Male | 302 | 304 | 606
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 817 | 795 | 1612
  Race: African American | 40 | 30 | 70
  Race: Other | 23 | 17 | 40
  Race: Missing | 117 | 169 | 286
Region of Enrollment [Number; unit: participants]
  United States | 997 | 1011 | 2008

OUTCOME MEASURES:

1. Primary Outcome: Do-Not-Resuscitate
Description: Percentage of residents with do-not-resuscitate orders documented in the electronic health record at end of follow-up, comparison between usual care and experimental arm
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Information
Number analyzed (Participants) | 997 | 1011
Participants | 144 | 136

2. Secondary Outcome: Do-Not-Hospitalize
Description: Percentage of residents in each arm with do-not-hospitalize or comfort care orders documented in the electronic health record at end of follow-up, comparison between usual care and experimental arm
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Information
Number analyzed (Participants) | 997 | 1011
Participants | 35 | 31

3. Secondary Outcome: Advance Care Planning Billing
Description: Percentage of residents in each arm with current procedural terminology billing code for advance care planning during follow-up based on Medicare claims data, comparison between usual care and experimental arm.
Time Frame: 4 months
Population: Only Medicare fee-for-service patients with linked claims data and complete Medicare coverage information were included in this analysis. Medicare Advantage patients were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Information
Number analyzed (Participants) | 743 | 770
Participants | 11 | 23

4. Secondary Outcome: Hospitalization
Description: Percentage of residents with any inpatient hospitalization during follow-up based on Medicare claims data (the MedPAR file), comparison between usual care and experimental arm.
Time Frame: 4 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Information
Number analyzed (Participants) | 743 | 770
Participants | 110 | 113

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the four months followup period for each resident
Arm/Group | Usual Care | Information
All-Cause Mortality (participants affected / at risk) | 35/1166 | 39/1198
Serious Adverse Events (participants affected / at risk) | 0/1166 | 0/1198
Other Adverse Events (participants affected / at risk) | 0/1166 | 0/1198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT04852055/Prot_SAP_000.pdf